CLINICAL TRIAL: NCT07302997
Title: A Single-Center, First-in-Human, Randomized, Controlled, Feasibility Study of a New Device for the Real-Time Continuous Monitoring of the Injection Pressure of Local Anesthetic in Subjects Undergoing Ultrasound-guided Peripheral Nerve Block: the Smart Needle Monitoring System Investigation
Brief Title: Real-Time Monitoring of the Injection Pressure During the Peripheral Nerve Block
Acronym: Smart Needle
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Principal Investigator, Dossi Roberto, MD, Ente Ospedaliero Cantonale, Bellinzona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025-D0048
Record Dates: First submitted 2025-11-27; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: No Condition; Real-time Monitoring of the Injection Pressure During Ultrasound-guided Axillary Block
Keywords: axillary block; injection pressure; real-time monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart Needle displaying (Experimental): The Smart Needle Monitoring System is used to perform the ultrasound-guided axillary block. The monitor connected to the Smart Needle will display real-time and record the injection pressure profile during the entire PNB procedure.
  The anesthesiologist will use the real-time visual feedback to maintain a low injection pressure profile (i.e., not higher than 15 psi) and avoid pressure peaks. The anesthesiologist can immediately stop the injection if there is a sudden increase in pressure, reposition the needle and start again, while always maintaining a low injection pressure profile
  Interventions: Device: Smart Needle Monitoring System
- Smart Needle flipped (Other): The Smart Needle Monitoring System is used to perform the ultrasound-guided axillary block. The monitor connected to the Smart Needle will be flipped allowing the recording of the injection pressure but not the real-time visualization by the anesthesiologist, who will perform the procedure as usual without a pressure visual feedback
  Interventions: Device: Smart Needle Monitoring System

INTERVENTIONS:
Device: Smart Needle Monitoring System — The Smart Needle Monitoring System is used to perform the ultrasound-guided axillary block. The monitor connected to the Smart Needle will display real-time and record the injection pressure profile during the entire PNB procedure

SUMMARY:
The goal of this clinical trial with medical device is to learn if the Smart Needle Monitoring System works to maintain a safe low injection pressure during a type of regional anaesthetic (Peripheral Nerve Block (PNB)) in patients due to undergo surgery below the elbow . It will also learn about the safety of the device and patients' perception of the quality of anesthesia.

Participants will:

* be operated locally according to standard clinical practice
* undergo post-anesthesia recovery and any neurologic symptoms or signs assessment on postoperative days 1 and 7

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* Age ≥ 18 years
* Scheduled for elective surgery below the elbow (e.g., hand surgery, distal radius surgery, forearm surgery) requiring an axillary block
* ASA physical status I-III
* Ability to understand the investigation
* Ability and willingness to follow and complete the procedures of the investigation

Exclusion Criteria:

* Contraindications to the axillary block (e.g., local infection)
* Refusal of locoregional anesthesia for the surgical procedure
* Pre-existing neurologic deficits in the operative extremity
* Body Mass Index ≥ 35 kg/m2
* Known allergy to local anesthetic (mepicavaine hydrochloride)
* Inability to comply with post-operative evaluations e.g. due to language problems, psychological disorders, dementia, etc. of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
proportion of injected nerves with at least one injection pressure peak in the investigational group compared to the standard (control) group | Perioperative
  The proportion of injected nerves with at least one injection pressure peak in the investigational group compared to the standard (control) group. A peak is defined as an injection pressure reaching a value above the threshold of 15 psi

SECONDARY OUTCOMES:
Success of the block | Perioperative
  Success of the block is defined as no conversion to general anesthesia (avoidance of rescue block, etc.)
Number of times of needle tip repositioning | Perioperative
  Number of times of needle tip repositioning, defined as the need to stop the ultrasound- guided PNB procedure to avoid excessive high pressure and reposition the needle tip
Total number of injection pressure peaks | Perioperative
  Total number of injection pressure peaks, i.e. raises of the injection pressure above the threshold of 15 psi, for each injected nerve
Quality of anesthesia from a patient's perspective | postoperative, 1 and 7 days after intervention
  Interview to the patient with 8 questions about quality of anesthesia from a patient's perspective in terms of pain, perception of needle movements and discomfort during the anesthesia procedure, and overall satisfaction; both Closed-ended questions and questions with scores 0 (worst) to 10 (best)

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Regionale di Bellinzona e Valli, EOC, Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided